CLINICAL TRIAL: NCT00313456
Title: A Phase I Study of the Oral Platinum Agent Satraplatin in Combination With Weekly Docetaxel
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decided to discontinue study drug development
Sponsor: Agennix (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAT1-05-09
Record Dates: First submitted 2006-04-10; First posted 2006-04-12 (Estimated); Last update posted 2012-05-10 (Estimated); Status verified 2012-05

CONDITIONS: Tumors; Prostate Cancer
MeSH Terms: conditions — Neoplasms; Prostatic Neoplasms | interventions — satraplatin

INTERVENTIONS:
Drug: Satraplatin — Satraplatin is an oral platinum analogue that has shown promising activity in multiple tumor settings. Satraplatin (40 to 80 mg/m2/day) will be administered orally on days 1 to 5 of a 21 day cycle.

SUMMARY:
This is a single-center, open-label (sequential-group dose-escalation dose-finding) phase I study of satraplatin and docetaxel in patients who have received prior chemotherapy regimens. Once the MTD is determined, an additional 6 patients, all with chemotherapy-naïve HRPC, will be enrolled. Once a recommended dose(s) (RD(s)) for phase 2 studies has/have been determined, 6 additional patients with chemotherapy-naïve HRPC will be enrolled at the RD to further evaluate safety and efficacy.

DETAILED DESCRIPTION:
RATIONALE:

Satraplatin is an oral platinum analog that is currently being evaluated in combination with prednisone in a phase III clinical trial in patients with HRPC who have progressed following one prior chemotherapy regimen.

Docetaxel is a taxane that is indicated for the treatment of patients with non-small cell lung, breast, and prostate cancers. Specifically, it was recently approved in combination with prednisone for the treatment of patients with hormone refractory prostate cancer (HRPC). Docetaxel administered every 3 weeks was associated with a survival advantage versus mitoxantrone. Docetaxel administered weekly showed an improvement in survival versus mitoxantrone that was not statistically significant. However, it was better tolerated than docetaxel administered every 3 weeks, with significantly less grade 3 and 4 toxicities, especially neutropenia. The combination of satraplatin and weekly docetaxel may be a feasible regimen for patients with chemotherapy-naïve HRPC and for patients with other malignancies for which these medications show activity.

OBJECTIVE:

The objective of this study is to determine the optimum doses for satraplatin and weekly docetaxel when the 2 drugs are given in combination.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven advanced solid tumors.
* 2 prior chemotherapy regimens.
* Age greater than or equal to 18 years.
* Eastern Cooperative Oncology Group performance status 0-1.
* Life expectancy greater than 3 months.
* At least 4 weeks between prior surgery or radiotherapy and enrollment.
* Adequate organ function as defined by the following criteria (must be obtained within 1 week of the first day of treatment):

Absolute neutrophil count ≥ 1500/µL. Hemoglobin ≥ 10.0 g/dl. Platelets ≥ 100,000/µL. Serum creatinine ≤ 1.5 upper limit of normal (ULN). Serum bilirubin ≤ ULN. AST/ALT ≤ 1.5 x the ULN.

* Patients must be able to swallow capsules.
* Patients must give written informed consent before study participation.
* No history of another cancer within the past 5 years (except basal or squamous cell carcinoma of the skin).
* No brain or leptomeningeal metastases.
* Female patients must not be pregnant or lactating and must be willing to practice contraception. Males must agree to contraceptive practices.

For HRPC cohort

* Patient must continue to be administered an LHRH agonist if they were receiving it at the time of screening for entry onto this protocol. Patients who have undergone bilateral orchiectomy do not need to be on LHRH agonists.
* Patient must be off of anti-androgen medications for ≥ 6 weeks.
* Patient must have castrate level of testosterone (< 50 ng/dL).
* Progressive HRPC as defined by one of the following:

  * Rising PSA
  * Sequential imaging studies
  * Clinical suspicion in the view of the treating physician

Exclusion Criteria:

* Patients who are unwilling to use contraception.
* Patients with a history of major gastrointestinal surgery.
* Pre-existing peripheral neuropathy > grade 1.
* Pre-existing edema > grade 1.
* Patients with hearing loss or tinnitus > grade 2.
* Prior RT to >25% of the bone marrow.
* Concomitant use of medications that inhibit cytochrome P450 3A4 (including aprepitant).
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational (utilized for non-FDA - approved indications and in the context of a research investigation).
* Patients who have not recovered (≥ grade 1) from the following toxicities of previous regimens before enrollment:

  * hematologic toxicities (parameters defined in protocol
  * fatigue
  * mucositis
  * nausea/vomiting/diarrhea.
* Uncontrolled intercurrent illness including, but not limited to, ongoing active infection, uncontrolled congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness that would limit compliance with study requirements.
* History of HIV or AIDS related illness.
* History of severe hypersensitivity reaction to docetaxel, polysorbate, or other drugs formulated with polysorbate 80.
* Evidence of concurrent second malignancy.
* History of bone marrow or major organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-03; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To assess the maximum tolerated dose (MTD) of satraplatin administered every 4 weeks in combination with docetaxel administered weekly (3 of 4 weeks) | 30 days

SECONDARY OUTCOMES:
To assess safety and tolerability (as per NCI-CTCAE version 3.0) | 30 days
To assess preliminary antitumor activity | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Petrone, MD, Study Director — GPC Biotech Inc.
Locations (1):
- Sarah Cannon Research Institute, Nashville, Tennessee, United States